CLINICAL TRIAL: NCT02484443
Title: A Phase 2 Study of Human-Mouse Chimeric Anti-disialoganglioside Monoclonal Antibody ch14.18 (Dinutuximab, NSC# 764038) in Combination With Sargramostim (GM-CSF) in Patients With Recurrent Osteosarcoma
Brief Title: Dinutuximab in Combination With Sargramostim in Treating Patients With Recurrent Osteosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-01001; NCI-2015-01001 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AOST1421; s16-00451; AOST1421 (Other: Children's Oncology Group); AOST1421 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2015-06-26; First posted 2015-06-29 (Estimated); Results first posted 2021-05-07 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Metastatic Malignant Neoplasm in the Lung; Metastatic Osteosarcoma; Recurrent Osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — dinutuximab; sargramostim; Colony-Stimulating Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (sargramostim and dinutuximab) (Experimental): Patients receive sargramostim SC QD on days 1-14 and dinutuximab IV over 10 hours on days 4-7 (dinutuximab infusion may be extended up to a total of 20 hours per day for anticipated toxicities). Treatment repeats every 28 days for up to 5 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Dinutuximab; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Biological: Sargramostim

INTERVENTIONS:
Biological: Dinutuximab — Given IV
  Other Names: Ch 14.18UTC; Ch14.18; Dinutuximab Beta; MOAB Ch14.18; monoclonal antibody Ch14.18; Qarziba; Unituxin
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Biological: Sargramostim — Given SC
  Other Names: 23-L-Leucinecolony-Stimulating Factor 2; DRG-0012; Leukine; Prokine; rhu GM-CFS; Sagramostim; Sargramostatin

SUMMARY:
This phase II trial studies how well dinutuximab works when given with sargramostim in treating patients with osteosarcoma that has come back after treatment (recurrent). Monoclonal antibodies, such as dinutuximab, may find tumor cells and help kill them. Sargramostim may help the body increase the amount of white blood cells it produces, which help the body fight off infections. Giving dinutuximab with sargramostim may work better and kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the disease control rate in patients with completely resected recurrent osteosarcoma treated with ch14.18 (dinutuximab) in combination with sargramostim (granulocyte-macrophage colony-stimulating factor [GM-CSF]) as compared to historical Children's Oncology Group (COG) experience.

SECONDARY OBJECTIVES:

I. To characterize the pharmacokinetics of ch14.18 (dinutuximab) in patients with recurrent osteosarcoma.

II. To determine the occurrence of unacceptable toxicity (UT) in patients with recurrent osteosarcoma treated with ch14.18 (dinutuximab) in combination with sargramostim.

III. To assess the relationship between probability of disease control and tumor ganglioside GD2 (GD2) expression.

TERTIARY OBJECTIVES:

I. To assess the relationship between probability of disease control and tumor GD2 expression.

II. To assess KIR and Fcgamma receptor (FcgammaR) genotypes, NKp30 isoforms and its circulating ligand, B7-H6, and their relationships to the probability of disease control.

III. To attempt banking of tumor samples for future research studies from patients enrolled on study who undergo biopsy or resection of suspected metastatic disease recurrence while on protocol therapy or during the evaluation period.

IV. To determine a descriptive profile of human anti-chimeric antibody (HACA) during immunotherapy.

V. To bank serial plasma samples for future studies of circulating tumor deoxyribonucleic acid (ctDNA) detection as a marker of disease progression and response.

OUTLINE:

Patients receive sargramostim subcutaneously (SC) once daily (QD) on days 1-14 and dinutuximab intravenously (IV) over 10 hours on days 4-7 (dinutuximab infusion may be extended up to a total of 20 hours per day for anticipated toxicities). Treatment repeats every 28 days for up to 5 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 8 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologic diagnosis of osteosarcoma at original diagnosis
* Patients must have had at least one episode of disease recurrence in the lungs without limitation on number of episodes of recurrence as long as they meet the following criteria:

  * Surgical resection of all possible sites of suspected pulmonary metastases in order to achieve a complete remission within 4 weeks prior to study enrollment**
  * Pathologic confirmation of metastases from at least one of the resected sites

    * For patients with bilateral pulmonary metastases, resection must be performed from both lungs and the study enrollment must be within 4 weeks from date of the last lung surgery
  * Note: If surgery related changes such as atelectasis are seen on the post-operative computed tomography (CT) scan, patients will remain eligible to enroll as long as the operating surgeon believes that all sites of metastases were resected; patients with positive microscopic margins will be eligible to enroll
* Patient must have adequate tumor specimen available for submission
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1 or 2; use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study

  * Myelosuppressive anti-cancer therapy: must not have been received within 2 weeks of study entry (4 weeks if prior nitrosourea)
  * Biologic (anti-neoplastic agent): at least 7 days since the completion of therapy with a biologic agent
  * Radiation therapy (RT): >= 2 weeks for local palliative radiation therapy (RT) (small port); >= 6 weeks must have elapsed if prior craniospinal RT or if >= 50% radiation of pelvis; >= 6 weeks must have elapsed if other substantial bone marrow (BM) radiation
  * Surgery: >= 2 weeks from last major surgery, including pulmonary metastasectomy, with the exclusion of a central line placement and core needle or small open biopsies
* Patient must not have received pegfilgrastim within 14 days of enrollment
* Patient must not have received filgrastim (G-CSF, Neupogen) within 7 days of enrollment
* Patient must not have received immune suppressants: corticosteroids (for other than allergic reactions and anaphylaxis), cyclosporine or tacrolimus within 7 days of enrollment

  * Note: the use of topical and/or inhalational steroids is allowed
* Total absolute phagocyte count (APC = [%neutrophils + %monocytes) x white blood cells [WBC]) is at least 1000/uL
* Platelet count >= 50,000/uL
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or
* A serum creatinine based on age/gender as follows:

  * 1 month to < 6 months: 0.4 (male) 0.4 (female)
  * 6 months to < 1 year: 0.5 (male), 0.5 (female)
  * 1 to < 2 years: 0.6 (male), 0.6 (female)
  * 2 to < 6 years: 0.8 (male), 0.8 (female)
  * 6 to < 10 years: 1 (male), 1 (female)
  * 10 to < 13 years: 1.2 (male), 1.2 (female)
  * 13 to < 16 years: 1.5 (male), 1.4 (female)
  * >= 16 years: 1.7 (male), 1.4 (female)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 110 U/L (for the purpose of this study, the ULN for SGPT is 45 U/L)
* Serum albumin >= 2 g/dL
* Baseline electrocardiogram (EKG) shows normal corrected QT interval (QTc) interval of =< 470 milliseconds (ms)
* Shortening fraction of >= 27% by echocardiogram, or
* Ejection fraction of >= 50% by radionuclide angiogram or echocardiogram
* No evidence of dyspnea at rest, no history of exercise intolerance, and a pulse oximetry > 94%
* Patient has no known history of seizure disorder
* Central nervous system (CNS) toxicity including peripheral neuropathy =< grade 2

Exclusion Criteria:

* Patients with distant bone metastases at original diagnosis or relapse (patients with only skip lesions will be eligible)
* Patients with concurrent local and pulmonary recurrence at the time of enrollment; note: patients who had local recurrence previously that has been treated and now present with an isolated pulmonary recurrence and meet the surgical resection criteria stated above will be eligible
* Patients with primary refractory disease with progression of the primary tumor on initial therapy
* Patients with CNS disease or other sites of extra-pulmonary metastases at the time of most recent episode of disease recurrence preceding enrollment
* Patients with a prior hypersensitivity reaction to sargramostim
* Patients who have received prior anti-GD2 therapy, including chimeric antigen receptor (CAR) T cells directed against GD2 antigen
* Female patients who are pregnant are ineligible
* Lactating females are not eligible unless they have agreed not to breastfeed their infants
* Female patients of childbearing potential are not eligible unless a negative pregnancy test result has been obtained
* Sexually active patients of reproductive potential are not eligible unless they have agreed to use an effective contraceptive method for the duration of their study participation; patients should maintain adequate contraception for a minimum of 2 months after the last dose of ch14.18 (dinutuximab)

Max Age: 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2016-02-04 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Hingorani, Principal Investigator — Children's Oncology Group
Locations (130):
- United States (111):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Beaumont Children's Hospital-Royal Oak, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Albany Medical Center, Albany, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (8):
  - John Hunter Children's Hospital, Hunter Regional Mail Centre, New South Wales
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Women's and Children's Hospital-Adelaide, North Adelaide, South Australia
  - Monash Medical Center-Clayton Campus, Clayton, Victoria
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (8):
  - Alberta Children's Hospital, Calgary, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - Children's Hospital, London, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch
- University Pediatric Hospital, San Juan, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Sargramostim and Dinutuximab)
Started | 41
Completed (Completion of planned therapy of Five Cycles and Disease Control Success (event-free for at least 12 months).) | 9
Not Completed | 32
Not completed — Lack of Efficacy | 28
Not completed — Physician Decision | 2
Not completed — Ineligible | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Sargramostim and Dinutuximab)
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 33
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 15 [7 to 26]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 27
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 37
  Australia | 2
  Canada | 1
  New Zealand | 1

OUTCOME MEASURES:

1. Primary Outcome: Disease Control
Description: Patients who can be confirmed to be free of detectable disease 12 months after enrollment, without intervening disease progression, will be considered to have demonstrated 12 month disease control. All other eligible patients will be considered not to have demonstrated 12 month disease control.
Time Frame: 12 months after study enrollment
Population: All eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Sargramostim and Dinutuximab)
Number analyzed (Participants) | 39
Participants | 11

2. Secondary Outcome: T 1/2 Alpha of the Serum Concentration of Dinutuximab
Description: T 1/2 alpha of the serum concentration of dinutuximab in days
Time Frame: Cycle 1 Day 4 and Day 7: pre-infusion, hour 4-6, end of infusion, 4-8 hours post infusion. Once between days 11-17. Cycle 2 Day 0 or 1
Population: Analysis population includes only patients for whom blood samples were submitted for pharmacokinetic analysis.
Measure: Median (Full Range); unit: days
Arm/Group | Treatment (Sargramostim and Dinutuximab)
Number analyzed (Participants) | 29
days | 0.8 [0.566 to 1.89]

3. Secondary Outcome: T 1/2 Beta of the Serum Concentration of Dinutuximab
Description: T 1/2 beta of the serum concentration of dinutuximab in days
Time Frame: as for outcome 2
Population: Analysis population includes only patients for whom blood samples were submitted for pharmacokinetic analysis.
Measure: Median (Full Range); unit: days
Arm/Group | Treatment (Sargramostim and Dinutuximab)
Number analyzed (Participants) | 29
days | 7.5 [7.25 to 7.86]

4. Secondary Outcome: Maximum of Concentration (Cmax) of the Serum Concentration Dinutuximab
Description: Cmax of the serum concentration dinutuximab as mg/L.
Time Frame: as for outcome 2
Population: Analysis population includes only patients for whom blood samples were submitted for pharmacokinetic analysis.
Measure: Median (Full Range); unit: mg/L
Arm/Group | Treatment (Sargramostim and Dinutuximab)
Number analyzed (Participants) | 29
mg/L | 18.4 [7.58 to 26.3]

5. Secondary Outcome: Area Under the Curve (AUC)0 to Infinity of Serum Dinutuximab
Description: (AUC)0 to infinity of serum dinutuximab in mg-h/L.
Time Frame: as for outcome 2
Population: Analysis population includes only patients for whom blood samples were submitted for pharmacokinetic analysis.
Measure: Median (Full Range); unit: mg-h/L
Arm/Group | Treatment (Sargramostim and Dinutuximab)
Number analyzed (Participants) | 29
mg-h/L | 2136 [904 to 2514]

6. Secondary Outcome: Number of Cycles Where an Unacceptable Toxicity as Defined in the Protocol Using The National Cancer Institute Common Terminology Criteria for Adverse Events Version 4 Was Observed
Description: The number of cycles where a dose-limiting toxicity was identified where dose-limiting toxicity is defined in the protocol using the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0. Occurrence of unacceptable toxicity as graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0, coded as present or absent, in each cycle received by eligible patients where all prescribed therapy for the cycle is received or the patient experiences unacceptable toxicity.
Time Frame: 5 cycles of protocol therapy planned as 140 days
Population: 39 patients were treated on protocol therapy. One hundred thirty-six cycles were reported for the analysis of dose limiting toxicity
Measure: Number; unit: cycles
Units Other Than Participants: Cycles
Arm/Group | Treatment (Sargramostim and Dinutuximab)
Number analyzed (Participants) | 39
Number analyzed (Cycles) | 136
cycles | 1

7. Other Pre Specified Outcome: Tumor GD2 Expression
Description: Archival tumor tissue will be assessed by immunohistochemistry to provide the level of GD2 expression in tissue as an integer between 0 and 3 with 0 indicating no GD2 expression and 3 indicating strong GD2 expression.
Time Frame: At study enrollment
Reporting Status: Not Posted

8. Other Pre Specified Outcome: KIR Genotype Analyses
Description: KIR mismatch will be assessed from the pre-treatment blood specimen as present or absent.
Time Frame: At enrollment
Reporting Status: Not Posted

9. Other Pre Specified Outcome: NKp30c Genotype Analyses
Description: Status of the immunosuppressive isoform of NKp30c KIR mismatch will be assessed from the pre-treatment blood specimen as present or absent.
Time Frame: At enrollment
Reporting Status: Not Posted

10. Other Pre Specified Outcome: FcgammaR Genotype Analyses
Description: FcgammaR genotype will be assessed from the pre-treatment blood specimen as H/R, R/R or H/H.
Time Frame: At enrollment
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Change in Circulating Ligand B7-H6 Levels
Description: The change in surface expression of ligand B7-H6 in terms of counts between the blood sample taken prior to the start of protocol therapy and the end of cycle 1 will be calculated. Patients who do not receive all prescribed protocol therapy during cycle 1 will not be evaluable for this outcome measure.
Time Frame: Cycle 1 of therapy planned to be 21 days
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Banking of Tumor Samples (Optional)
Description: Individual statistical plans will be developed for future studies answering a specific question using these banked tumor specimens.
Time Frame: 5 cycles of protocol therapy planned as 140 days
Reporting Status: Not Posted

13. Other Pre Specified Outcome: HACA Titer
Description: HACA titer will be determined in each blood sample provided to the HACA reference laboratory.
Time Frame: At enrollment, at the start of each cycle of therapy and within 30 days of the end of cycle 5
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Circulating Tumor Deoxyribonucleic Acid Detection
Description: Statistical considerations for specific future studies will be provided.
Time Frame: 5 cycles of protocol therapy planned as 140 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Through completion protocol therapy planned as 140 days after study enrollment
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Arm/Group | Treatment (Sargramostim and Dinutuximab)
All-Cause Mortality (participants affected / at risk) | 15/39
Serious Adverse Events (participants affected / at risk) | 12/39
Other Adverse Events (participants affected / at risk) | 28/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Sargramostim and Dinutuximab) (N=39)
Blurred vision (Eye disorders) | 2 (2)
Eye disorders - Other, specify (Eye disorders) | 1 (1)
Photophobia (Eye disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Fever (General disorders) | 1 (1)
Sudden death NOS (General disorders) | 1 (1)
Serum sickness (Immune system disorders) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Sargramostim and Dinutuximab) (N=39)
Abdominal pain (Gastrointestinal disorders) | 8 (8)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 7 (7)
Allergic reaction (Immune system disorders) | 5 (5)
Cytokine release syndrome (Immune system disorders) | 1 (1)
Serum sickness (Immune system disorders) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
GGT increased (Investigations) | 2 (2)
Lymphocyte count decreased (Investigations) | 3 (3)
Neutrophil count decreased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 1 (1)
Urine output decreased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
Capillary leak syndrome (Vascular disorders) | 8 (8)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-22): https://cdn.clinicaltrials.gov/large-docs/43/NCT02484443/Prot_SAP_000.pdf